CLINICAL TRIAL: NCT07071259
Title: Study of the Correlation Between Cortical Excitability and Cytoarchitectonics of Prefrontal Cortex in Healthy Adult Participants, Using Transcranial Magnetic Stimulation Coupled to EEG and High-field MRI
Acronym: FrontalProbe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C23-43; 2024-A02244-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants; Magnetic Stimulation; MRI; EEG; Dorsolateral Prefrontal Cortex; rTMS Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of data during stimulation of 3 DLPFC subregions (Active Comparator)
  Interventions: Other: TMS Stimulation

INTERVENTIONS:
Other: TMS Stimulation — For the TMS session, participants will be positioned on a chair, in a seated position. They will be equipped with an EEG cap 64 active electrodes, using gel to ensure good measurements of brain activation, and a sensor on the forehead to measure the location of the head in space for the neuronavigation system. They will also wear headphones generating white noise to mask the TMS coil noise. Preparation time for the EEG acquisitions is estimated at 30 min. The TMS coil will be shaped in 8 for good spatial resolution. It will be positioned on the participant's head using a robot (approved medical CE) allowing good targeting accuracy and stability during the experiment. The stimulation target will be defined beforehand on the participant's MRI, and the robot will read this information to position itself.

SUMMARY:
Repeated transcranial magnetic stimulation (rTMS) is mainly used to treat mood disorders by addressing differences in brain function, particularly in the dorsolateral prefrontal cortex (DLPFC), which affects emotions and executive functions. The therapy aims to enhance the left DLPFC or suppress the right. It has been approved for severe major depression in several countries (Canada and Israel since 2002, USA since 2008) and is in the process of being validated in Europe but is not yet reimbursed in France. due to variable results from one study to another and lack of standardization issues.

In a previous study, by recording electroencephalographic (EEG) rhythms before and after rTMS treatment of the DLPFC, the investigators showed on a small cohort of patients (n=17) with major or bipolar depression, that the responder patients showed higher EEG theta rhythms in the DLPFC but also and especially in parietal regions. This suggests that the DLPFC is part of the fronto-parietal central executive network (CEN), which is important for working memory and cognitive control. The CEN is not well connected in severe resistant depression, possibly leading to negative emotional bias. The rTMS cure of DLPFC can be interpreted as improving depressive symptoms through the normalization of the CEN by increasing DLPFC excitability and its downward connectivity. However experimental and clinical evidence for this mechanism, among others, is still to be demonstrated, and remission rates of rTMS from DLPFC in drug-resistant depression are still low (20-40%).

To improve these response rates to rTMS in DLPFC, it is essential to continue research aimed at improving clinical practices through a better knowledge of the functional neuroanatomy and mechanisms of action of rTMS. This will require the definition of biomarkers allowing in particular to better target the DLPFC, this structure beeing indeed relatively poorly defined on the neuroanatomical level (large portion of the medial frontal gyrus). To this end, the investigators have set up a collaborative research program with Dr. Corey Keller, psychiatrist at Stanford University USA, which was jointly funded in 2022 by the Agence Nationale pour la Recherche (ANR) and the National Institute of Health (NIH) - FrontalProbe project "Probing the dorsolateral prefrontal cortex and central executive network for improving neuromodulation in depression". The ultimate aim of this project is to develop and test different strategies for targeting the DLPFC in the rTMS treatment of pharmaco-resistant depressive patients, following the fundamental neuroanatomical and pathophysiological hypothesis that patients will respond better to therapy if their CEN network is better modulated. This clinical trial will take place in Stanford, USA, in the years 2025-2026. Previously, the investigators are working on the development of methodological strategies aimed at preferentially activating, in a personalized way, the part of the DLPFC that projects onto the PPC. This is the subject of the present protocol, which aims to identify this subpart of the DLPFC to be targeted as a priority for modulating the CEN, through neuroanatomical measurements with high-field MRI and cortical excitability by TMS-EEG in healthy subjects. To this end, the investigators will use a small cohort of healthy subjects who will have one multimodal MRI acquisition session of at 7T and one TMS-EEG session. The 7T MRI data, acquired at the Centre de Résonance Magnétique en Biologie et Médecine (CRMBM), will be used to obtain anatomical markers of the DLPFC. TMS-EEG data, acquired at the Institut de Neurosciences de Systèmes (INS), will be used for cortical excitability measurements of the DLPFC and its projection sites, notably the PPC. At this stage, no data exchange is planned with our American partners.

Firstly, the processing of MRI data will include segmentation of gray and white matter, reconstruction of the cortical surface and estimation of the different cortical layers, mainly by monitoring variations in the T1 parameter along the cortical mantle. Other MRI parameters will also be acquired to maximize the specificity of the segmentation of the DLPFC into sub-regions, firstly by identifying the part of the DLPFC that connects preferentially to the PPC using the reconstruction of fiber bundles from diffusion MRI and functional resting MRI. Secondly, during TMS-EEG acquisitions, participants will be stimulated in 3 sub-regions of the DLPFC. For each target, the analyses of the EEG data will focus on quantifying connectivity with the PPC as well as their spectral signature, which is possibly an indirect reflection of the neuronal composition of the stimulated regions.

Correlation of 7T MRI and TMS-EEG data will help set optimal DLPFC targeting criteria for PPC activation. The aim is to create an MRI-based targeting procedure for clinical practice. In this sense, TMS-EEG will serve as validation of MRI markers.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 to 35
* People affiliated with a social security scheme or beneficiary of such a scheme
* People who have signed the informed consent
* Right-handed people
* People with a body mass index between 18 and 26
* People able to abstain from alcohol for 24 hours prior to the experiment
* People able to remain perfectly still for 15 minutes straight, and able to have reduced mobility for 3 hours
* People able to of not using narcotics (marijuana, cocaine, ecstasy, MDMA, ketamine, etc.) during the 15 days preceeding the experiment.
* Conducting a pregnancy test before inclusion for women of childbearing age and when the research is conducted over a long period, at a frequency adapted to the gaze of the research acts
* Effective contraception for women of childbearing potential

Exclusion Criteria:

* Pregnant, parturient, or breastfeeding
* Protected adults
* Minors
* People staying in a healthcare or social institution
* People in an emergency situation
* People deprived of their liberty
* People with the usual contraindications to MRI

  * Ferromagnetic surgical clips, ocular implants, metallic foreign bodies intraocularly or in the nervous system, implants or metallic objects susceptible to concentrate the radio frequency field, cochlear implants, brain stimulator or cardiac pacemaker, presence of a craniotomy scar, agitation
  * Claustrophobia
  * Large, black tattoo close to the orofacial area
* People not wishing to be informed of abnormalities discovered at the MRI
* People with a history of epilepsy or suffering from epilepsy
* Individuals whose parents, children, siblings, or parents have a history of epilepsy
* People with known neurological and/or psychiatric disorders with past and/or current medical treatment, or drug addiction
* Staff with a hierarchical link to the investigators

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of TMS-EEG session | between Day 1 and Day 30
  Participants will be stimulated in three subregions of the DLPFC. The TEP (Transcranial Evoked Potential) will be reconstructed at the parietal and frontal cortical areas using "Minimum Norm" EEG source reconstruction algorithms as provided in the Brainstorm software (https://neuroimage.usc.edu/brainstorm/Tutorials/SourceEstimation).

SECONDARY OUTCOMES:
Multimodal MRI examination at 7T | One or more days before the TMS-EEG session
  Diffusion MRI scans will be analyzed using tractography methods (e.g. MRTrix, Connectomist, FSL) to reconstruct fiber bundles at the individual level between segmented prefrontal and parietal areas.